CLINICAL TRIAL: NCT04040062
Title: Pilot Study: Evaluating the Feasibility of Repetitive Transcranial Magnetic Stimulation Treatment Delivered at Individual-based, SCC-determined Frequency in Subjects Suffering From Major Depressive Disorder
Brief Title: Spectral Correlation Coefficient-based TMS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Director of UCLA Neuromodulation, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0758; NCT04166864 (obsolete NCT alias)
Record Dates: First submitted 2019-07-08; First posted 2019-07-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: We will identify the participant's individual spectral correlation coefficient (SCC) by stimulation with 68 different stimulation pulse trains of 40 pulses each at frequencies ranging between 3 and 20 Hz in steps of 0.25 Hz, plus intermittent theta burst (iTBS) stimulation, in randomized order. We will then select the frequency with the largest connectivity density (strong and focal connectivity increase within the fronto-parietal control network) in the range of 3 and 20 Hz as the optimal individual stimulation density and treat the participants at this optimal Hz for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCC (Experimental): Subjects will be treated according to their frequency response pattern which may show one or more distinct frequencies of stimulation that generated increased SCC
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain to improve symptoms of depression. Using pulsed magnetic fields, transcranial magnetic stimulation therapy stimulates the part of the brain thought to be involved with mood regulation. These magnetic fields do not directly affect the whole brain; they only reach about 2-3 centimeters into the brain directly beneath the treatment coil.As these magnetic fields move into the brain, they produce very small electrical currents. These electrical currents activate cells within the brain, causing them to rewire, a process called neuroplasticity.

SUMMARY:
This study will analyze the feasibility, safety, and tolerability of administering repetitive Transcranial magnetic stimulation(TMS) at frequencies other than standard 10 Hz. This study will enroll 50 subjects who will undergo one quantitative electroencephalograph, one TMS procedure to determine the appropriate frequency and intensity for treatment, weekly mood/symptom assessments, and up to 30 TMS treatments. Subjects will be asked to participate for up to 6 weeks.

DETAILED DESCRIPTION:
The therapeutic benefit of repetitive Transcranial Magnetic Stimulation (rTMS) for the treatment of Major Depressive Disorder (MDD) is thought to depend upon engagement of brain functional networks (FNs). Engagement is dependent upon an interaction between the rTMS stimulation frequency and the preferred oscillatory frequency of the target network for that individual. We report here on a novel method to interrogate the left dorsolateral prefrontal cortex (DLPFC) treatment target to identify the optimal frequency for engagement of the frontoparietal control network (FCN) for each individual. 23 subjects with MDD were stimulated with 40 pulse rTMS trains at frequencies varying from 3-17 Hz at 0.2 Hz increments, plus a separate intermittent theta burst (iTBS) stimulation, for a total of 70 frequency interrogations. FN engagement was assessed using continuous high-density array TMS-EEG recordings and measurement of the change in the density of the spectral correlation coefficient (SCC) between left DLPFC and other brain areas following each interrogation. All subjects had one or more frequency bands that showed high SCC values across multiple FNs, regardless of the frequency of interrogation. Those subjects who showed clinical response to 10 Hz rTMS showed increases in SCCD over FCN connections across in response to 10 Hz interrogation, but not in response to interrogation in other bands. There was a strong association between the increase in SCCD in FCN and degree of improvement in depressive symptoms after both 2 and 6 weeks of treatment. These findings suggest that SCC density may be useful for identifying rTMS stimulation frequencies that are associated with therapeutic benefit in MDD. This study will examine the feasibility using these findings to determine if SCC-determined rTMS treatment can benefit subjects with Major Depressive Disorder.

INTRODUCTION AND RATIONALE

Repetitive Transcranial Magnetic Stimulation (rTMS) has been reported to relieve symptoms of Major Depressive Disorder (MDD) when administered at a number of different stimulation frequencies: 1, 5, 10, 15, 18, and 50 Hz (theta burst stimulation, or TBS) all have reported to provide clinical benefit. It is difficult to compare the efficacy of these different frequencies of stimulation because of differences in study design and limitations of sample size, but there is significant evidence of efficacy for each of these frequencies when applied to one or more stimulation targets.1 There have not been head-to-head studies to compare different stimulation frequencies in individual subjects to determine whether individuals have similar clinical responses to more than one frequency of stimulation.

One feature that is shared by all frequencies of rTMS is that while stimulation is ongoing, both neuronal spiking and ongoing oscillations are synchronized to the frequency of stimulation (Fröhlich and McCormick, 2010 ; Thut et al., 2011 ). This modulation of cerebral oscillatory activity is hypothesized to underlie the therapeutic effects of rTMS for MDD. , Entrainment of brain oscillations has been shown to modify brain activity in a variety of functional networks (FNs), with changes in oscillations associated with alterations in task performance, local oscillatory activity, connectivity patterns and in the case of motor networks, corticospinal coupling.

Different frequencies of rTMS stimulation have distinct effects on FN engagement and task performance. These differential effects are consistent with the fact that FNs have one or more preferred resonant frequencies that mediate connectivity both within and across networks (Hacker et al., 2017 , , , The effects of rTMS stimulation depends upon the interaction between the frequency of stimulation and the ongoing oscillatory activity of the target FN(s): the oscillatory pattern of the specific brain region being stimulated (as measured with electroencephalography [EEG]) is a major determinant of rTMS engagement with the associated FN(s)3, and the effects on network performance.

The frontoparietal control network (FCN) is of particular interest in MDD because it is dysregulated in MDD, with the degree of dysfunction related to severity of depressive symptoms. The most commonly used neuroanatomic rTMS stimulation target is left dorsolateral prefrontal cortex (DLPFC), which is a critical hub of the FCN. Furthermore, the FCN plays a crucial role integrating the function of multiple other FNs. , , 10 Hz is the most commonly rTMS stimulation used to stimulate the left DLPFC target, but it has not been established that this frequency is optimal for engaging the FCN. Multiple stimulation frequencies have differential effects on the FCN, changing FCN interactions with default mode network (DMN) from excitatory to inhibitory. This finding is consistent with the fact that adjusting the frequency of stimulation affects which nodes within a single FN are engaged, , the extent to which rTMS stimulation engages local vs. distant network modules, and selectively alters the engagement between a FN and an affiliated brain region. FCN connectivity is known to be mediated by multiple frequencies ranging from 2 Hz (delta band) though 20 Hz (beta band) (Johnson et al., 2019 ; Lopez et al., 2019 ; Cooper et al., 2015 ; 18).

The present study was performed to determine whether it was possible to identify differential effects of rTMS treatment frequency on engagement of the FCN during rTMS treatment of MDD, through examination of frequency coupling across a broad spectrum of stimulation frequencies within the FCN. It was recently reported that changes in whole-brain spectral connectivity in the frequency band (alpha spectral correlation, or SC) from pre- to post- the first session of 10 Hz rTMS applied to left DLPFC predicted outcome from a course of 30 rTMS treatments. In the current study, we examined spectral correlation across a broad frequency spectrum following a series of rTMS "interrogations" ranging from 3 Hz to TBS. This allowed us to generate a spectral correlation coefficient (SCC) across this frequency spectrum and determine which frequencies of stimulation would lead to increased SCC within the FCN. This study hypothesizes that: 1) each subject's frequency response pattern would show one or more distinct frequencies of stimulation that generated increased SCC; 2) these frequency response patterns would differ across subjects, but be highly reproducible within subjects over a course of rTMS treatment; and, 3) those subjects with concentrated increases in FCN SCC (increased SCC density) following 10 Hz interrogation would be more likely to show clinical response to 10 Hz rTMS treatment.

STUDY OBJECTIVE

The primary objective of this study is to demonstrate feasibility of rTMS treatment for depression at stimulation frequencies other than 10 Hz. Objectives:

1. to determine if each subject's frequency response pattern shows one or more distinct frequencies of stimulation that generated increased SCC;
2. to determine if these frequency response patterns differ across subjects; and,
3. To gather pilot data for an extramural funding application to investigate the efficacy of rTMS treatment at individualized stimulation frequencies as an alternative to the standard 10 Hz protocol.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be over between 18-65 years of age.
* Must have confirmed diagnosis of severe Major Depressive Disorder (single or recurrent episode).
* Failure to respond to a minimum of 4 trials of antidepressant medication
* Failure to respond from at least two different agent classes
* Accompanied by at least two evidence-based augmentation therapies (Benzodiazepines do not count).
* Must have a trial of psychotherapy known to be effective in the treatment of MDD of an adequate frequency and duration.
* Subjects are willing and able to adhere to the treatment schedule and required study visits

Exclusion Criteria:

* Are mentally or legally incapacitated, unable to give informed consent
* Have an infection or poor skin condition over the scalp where the device will be positioned
* Have increased risk of seizure because of family history, stroke, or currently use medications that lead to increased risk for seizure
* Diagnosis of acute or chronic psychotic symptoms or disorders (such as schizophrenia, schizophreniform or schizoaffective disorder) in the current depressive episode.
* Neurological conditions that include epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, having a history of repetitive or severe head trauma, or with primary or secondary tumors in the central nervous system.
* Presence of an implanted magnetic-sensitive medical device located less than or equal to 30 centimeters from the transcranial magnetic stimulation magnetic coil or other implanted metal items, including but not limited to a cochlear implant, implanted cardioverter defibrillator, pacemaker, vagus nerve stimulator, or metal aneurysm clips or coils, staples, or stents.

(Note: Dental amalgam fillings are not affected by the magnetic field and are acceptable for use with transcranial magnetic stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Inventory of Depressive Symptoms- Self report | Weekly
  This survey is designed to assess the severity of depressive symptoms. The IDS assess all the criterion symptom domains designated by the American PsychiatryAssociation Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV) (APA1994) to diagnose a major depressive episode. These assessments can be used to screen fordepression, although they have been used predominantly as measures of symptom severity. The seven day period prior to assessment is the usual time frame for assessing symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided